CLINICAL TRIAL: NCT04861662
Title: Clinical and Radiographic Evaluation of the Effect of Keratinized Mucosa on Peri-implant Health
Brief Title: Effect of Keratinized Mucosa on Peri-implant Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Asst. Prof. Ezgi GÜRBÜZ, DDS, Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Keratinized Mucosa; Dental Implant; Free Gingival Graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Keratinized Mucosa Sufficient (KMS) (No Intervention): Implants exhibiting the width of keratinized mucosa (KM) ≥2 mm at the midbuccal aspect
- Keratinized Mucosa Deficient (KMD) (No Intervention): Implants exhibiting KM<2 mm at the midbuccal aspect
- Free Gingival Graft (FGG) (Experimental): Implants with KM<2 mm initially and having surgically increased keratinized mucosa with free gingival graft after prothesis delivery
  Interventions: Procedure: Free gingival graft procedure

INTERVENTIONS:
Procedure: Free gingival graft procedure — Free gingival graft procedure applied to implants with KM<2 mm to increase the width of keratinized mucosa surrounding them
  Arms: Free Gingival Graft (FGG)

SUMMARY:
The aim of this clinical study is to evaluate the significance of keratinized mucosa and to investigate the influence of free gingival graft procedure on peri-implant health status in patients after prothesis delivery.

DETAILED DESCRIPTION:
The study will be conducted in Faculty of Dentistry, Kutahya Health Sciences University . The patients who applied to the Department of Periodontology, received dental implant treatment, and required routine follow-up for the maintenance of peri-implant health will be included. Clinical and radiographic examinations will be performed at baseline (prothesis delivery) and at the end of the 3rd, 6th month, 1st year following the prosthetic loading. During clinical examination probing depth (PD), modified plaque index (mPI) and modified bleeding index (mBI) measurements will be evaluated with the Williams periodontal probe. These measurements will be taken at four points of the implant (mid-buccal, mesio-buccal, disto-buccal and mid-lingual) and these four measurements will be averaged for each implant. In addition, the amount of keratinized mucosa (KM) in the implant sites will be evaluated by measuring the mucosal margin and mucogingival junction on the vestibular surface with the same probe. After clinical examination, a periapical radiograph will be taken using a parallel technique to determine marginal bone loss surrounding the implant. The distance between the implant neck and the most coronal part of the alveolar crest will be measured on the mesial and distal surfaces for each implant on the obtained radiographs and the average of the two measurements will be taken. The parameters checked during clinical and radiographic examination will be compared between patients with or without keratinized mucosa and whose keratinized mucosa has been increased by free gingival graft.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Having dental implant treatment and prosthetic restoration
* Not having received bone augmentation treatment at the implant site
* To comply with maintenance controls after dental implant treatment

Exclusion Criteria:

* Pregnancy
* Having used systemic antibiotics within 6 weeks prior to the start of the study
* Having a disease that affects bone and soft tissue metabolism, such as hyperthyroidism, hyperparathyroidism, and uncontrolled diabetes mellitus
* Using drugs that cause immunosuppression
* Using a medicine that affects bone metabolism, such as a bisphosphonate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | Baseline, 3rd month, 6th month and 1st year
  Change of marginal bone loss measured from periapical radiographs

SECONDARY OUTCOMES:
Modified bleeding index | Baseline, 3rd month, 6th month and 1st year
  Parameter showing peri-implant mucosa inflammation
Probing depth | Baseline, 3rd month, 6th month and 1st year
  The depth of peri-implant sulcus in millimeters
Modified plaque index | Baseline, 3rd month, 6th month and 1st year
  Parameter showing oral hygiene performance

CONTACTS AND LOCATIONS:
Overall Officials: Melike Başaran, Principal Investigator — melike_basaran@ksbu.edu.tr
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)